CLINICAL TRIAL: NCT00968877
Title: Vitamin D and Chronic Renal Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Nephrological department, Peter Marckmann
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vita-D3
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2009-12

CONDITIONS: Vitamin D Deficiency; Chronic Renal Insufficiency
Keywords: Renal Insufficiency; Cholecalciferol; Kidney Disease; Kidney Failure; Vitamin D; Vitamin D Deficiency; Vitamin D3
MeSH Terms: conditions — Vitamin D Deficiency; Renal Insufficiency, Chronic; Renal Insufficiency; Kidney Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Active Comparator)
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — capsule 40 000 IU (p.o.) once per week, in 8 weeks.
  Other Names: Dekristol

SUMMARY:
Purpose of this study is to investigate the effect of treatment with vitamin D3 (cholecalciferol) compared with placebo in a trial including chronic kidney disease patients with vitamin D deficiency.

DETAILED DESCRIPTION:
Most patients with chronic renal insufficiency have vitamin D deficiency. It is still not common practice among nephrologists to monitor and correct vitamin D deficiency of chronic kidney disease (CKD) patients, because it is widely believed that any vitamin D deficiency associated with calcium-phosphate disturbances is better treated with activated vitamin D.

However, correction of vitamin D deficiency with native vitamin D seems to have numerous favorable effects not only related to the renal and intestinal handling of calcium and phosphate. It may have beneficial effects on bone and vascular health, the immune system and physical performance that are not obtained with active vitamin D treatment.

We are therefore planning a randomized, placebo-controlled, intervention study of 8 weeks' duration in which vitamin D3 supplementation (40 000 IE per week in one capsule) is compared with placebo in a trial including 120 CKD patients with vitamin D deficiency. Multiple biological variables are monitored in order to assess any effect on the biological systems of interest.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease (CKD 3-5 amd renal transplanted patients)
* Age > 18 years
* Vitamin D insufficiency or deficiency (25-OHD < 50 nmol/l, 3 months before project start)

Exclusion Criteria:

* Treatment with vitamin D2/D3 (dose more than 10000 IU within the last 3 months)
* Hypercalcaemia (ca++ > 1,35 mmol/l more than 4 weeks despite missing intake of calcium containing preparations and activated vitamin D)
* Uncontrolled hyperphosphataemia (s-phosphate > 2,2 mmol/l)
* Sarcoidosis
* Malignant disease
* Psychotic disorders
* Pregnancy and lactation women
* Allergy to soya and peanut

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Calcium phosphate associated metabolites, bone markers, endothelial markers, inflammation muscle function, pulse wave velocity test | 8 weeks

SECONDARY OUTCOMES:
Health questionnaire | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Marckmann, Prof, DMSc, Study Director — Nephrological department, Odense University Hospital